CLINICAL TRIAL: NCT02106312
Title: Dose Reduction of Preoperative Radiotherapy in Myxoid Liposarcomas
Acronym: DOREMY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N10DMY; 2588 (Other: Nederlands trial register)
Record Dates: First submitted 2014-03-06; First posted 2014-04-08 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2020-06

CONDITIONS: Myxoid Liposarcoma of Soft Tissue
Keywords: Radiotherapy; Myxoid liposarcoma; Soft tissue sarcoma
MeSH Terms: conditions — Liposarcoma, Myxoid; Sarcoma | interventions — cytochrome C synthetase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation (Other): Dose reduction of preoperative radiotherapy in MLS from 50 Gy to 36 GY.
  Interventions: Radiation: dose reduction of preoperative radiotherapy in MLS

INTERVENTIONS:
Radiation: dose reduction of preoperative radiotherapy in MLS — A: The primary sarcoma in case of non-metastatic disease for management is with curative intent (regime to be chosen=18 x 2 Gy) B: In case of oligometastatic patients, the metastasis may also be irradiated to a dose of 36 Gy in order to postpone the time interval to next systemic chemotherapy. These patients are usually not operated upon and the total dose may also be reached in 12 times 3 Gy, for convenience purposes.

SUMMARY:
To study the feasibility of reducing the dose of preoperative radiotherapy in MLS (Myxoid Liposarcomas) from 50 Gy to 36 Gy while maintaining comparable clinicopathological responses.

DETAILED DESCRIPTION:
* A Bayesian approach is considered for the analysis of this trial. The aim is to provide a stopping rule for inefficacy of the new dose.
* Two aspects are important to elucidate the mechanism of this treatment: dynamic investigations of perfusion and vasculature. Apart from participation to the dose reduction paragraphs of this study, patients will be also asked to undergo, at clinically relevant dose points, dynamic contrast enhanced (DEC) MRI scans and separately tumor biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Age above or equal to 18 years
2. Biopsy proven MLS (including the reciprocal chromosomal translocation t(12;16)(q13;p11); A the primary sarcoma in case of non-metastatic disease for management is with curative intent (regimen to be chosen = 18 x 2 GY) B in case of oligometastatic patients, the metastasis may also be irradiated to a dose of 36 GY in order to postpone the time interval to next systemic chemotherapy. These patients are usually not operated upon and the total dose may also be reached in 12 times 3 Gy, for convenience purposes (see paragraph 10 for radiobiological considerations).
3. ECOG (Eastern Cooperative Oncology Group) PS (Performance Status) 0-2
4. Patients must be able (physically, mentally and socially) to complete a series of RT, followed by an observation period of 4-6 weeks and undergo surgery.
5. Written informed consent

Exclusion Criteria:

1. Prior radiotherapy to the target area.
2. Anticoagulant medication of any kind; especially Ascal®(and derivates), coumarines (Sintrom® and Marcoumar®), all heparin and heparin-like formulations. (Note: this exclusion criterion only applies for patients consenting to the translational research part of the study; patients on anticoagulant medication as described above may take part in the dose reduction part of the study, but the repeat biopsies may not be taken.)
3. Pregnancy -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-12-15 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
The Pathological description of the percentage pathological responses after reduced RT (radiotherapy) dose from (conventionally) 25 x 2 Gy to 18 x 2 Gy (in the current study) | The percentage of pathological responses will be pathologically assessed on the resection specimen; this procedure will take on average 7-10 working days. After surgery, patients will be followed up to 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Rick Haas, MD,PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (12):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Harvard Cancer Center, Boston, Massachusetts
- University Hospital Aarhus, Aarhus, Denmark
- Netherlands (6):
  - The Netherlands Cancer Institute, Amsterdam, North Holland
  - Academisch Medisch centrum, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Leids Universitair Medisch Centrum, Leiden
  - Maastro Clinic, Maastricht
  - Radboud umc, Nijmegen
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
- Royal Marsden Hospital, London, United Kingdom

REFERENCES:
- [Derived] Lansu J, Bovee JVMG, Braam P, van Boven H, Flucke U, Bonenkamp JJ, Miah AB, Zaidi SH, Thway K, Bruland OS, Baldini EH, Jebsen NL, Scholten AN, van den Ende PLA, Krol ADG, Ubbels JF, van der Hage JA, van Werkhoven E, Klomp HM, van der Graaf WTA, van Coevorden F, Schrage Y, van Houdt WJ, Haas RL. Dose Reduction of Preoperative Radiotherapy in Myxoid Liposarcoma: A Nonrandomized Controlled Trial. JAMA Oncol. 2021 Jan 1;7(1):e205865. doi: 10.1001/jamaoncol.2020.5865. Epub 2021 Jan 21. PMID 33180100